CLINICAL TRIAL: NCT03847831
Title: Postprimary Active School Flag Feasibility
Brief Title: Feasibility Study of the Pilot Post-primary Active School Flag (PPASF) Program
Acronym: PPASF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Principal Investigator, Kwok Ng, Healthy Ireland Demonstration Project Project Manager, University of Limerick
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Postprimary Active School Flag
Record Dates: First submitted 2019-02-12; First posted 2019-02-20 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Physical Activity; Health Behavior; Health Knowledge, Attitudes, Practice; Educational Problems
Keywords: whole-school; health promotion
MeSH Terms: conditions — Motor Activity; Health Behavior; Behavior

STUDY DESIGN:
Intervention Model Description: Non-randomised single-group at school level pilot study.
Masking Description: This is a pilot study of schools enrolled into a program. The students and teachers in the schools are the subjects exposed to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PPASF Group (Experimental): Schools enrolled in the post primary active school flag program. All 17 elements are included. Feasibility is measured of the 17 elements.
  Student representatives are selected to have accelerometer, physical health measures and perceived health collected for feasibility purposes.
  Interventions: Behavioral: Active School Flag Program

INTERVENTIONS:
Behavioral: Active School Flag Program — Schools enrolled in the program take part in the 17 actions described in the PPASF.

SUMMARY:
The Feasibility of the post-primary Active School Flag (PPASF) programme. The PPASF is an initative from the Department of Education and Skills in a whole-school program to increase physical activity opportunities involving the students in second level education schools in Ireland. Various actors involved in the process include admin, teachers, and students to create more physical activity opportunities for the students in the school. Process evaluation and fidelity of the program are carried out during the year long process for certificate and two years for achieving the flag. Results of this study will inform the design and implementation of the PPASF in a national roll out across Irish second level education schools.

DETAILED DESCRIPTION:
This is a feasibility study of the post-primary Active School Flag (PPASF) programme. Schools in Ireland that meet the eligibility criteria of; 1) second level education school, 2) has not already achieved the Active School Flag, 3) volunteered to be in the study were selected to take part in this pilot study. Schools not in the programme were matched to provide a comparison data set.

Schools involved in the study are given resources to support the year long program so the school may achieve the PPASF certificate. To achieve the certificate, the schools needed to complete 17 tasks throughout the school year; 1) a staff slideshow, 2) an PPASF team slideshow, 3) class time slideshow 4) PPASF training day, 5) an PPASF awareness week (towards the beginning of the year), 6) website showcase, 7) PPASF whole school questionnaire, 8) PPASF launch event, 9) PPASF action plan, 10) 'Did You Know?' campaign, 11) PA module as part of Social, personal and health education (SPHE) subject for junior cycle students, 12) Active School WALKWAY, 13) Community Mapping of extra curriculum activities, 14) Community Event, 5) Active School Week, 16) PPASF accreditation visit, and 17) school PA space audits.

The PPASF is part of the developing Healthy Ireland Demonstration Project, and the feasibility to collect data in the form of accelerometers, physical health measures and self-perceptions of health are also included in the feasilibility study.

The feasibility study will be monitored quantitatively through a custom design fidelity check list, and in depth process evaluation that includes qualitative methods such as one to one interviews and focus group interviews throughout the academic year.

The secondary outcomes are based on the hypotheses that 1) intervention schools will have more physical activity opportunities and thus 2) more physically active students, especially during the school day. Furthermore, there would be 3) a decrease in sitting time, 4) positive associations between academic related behaviours with physical activity behaviours, 5) and no increase in BMI.

ELIGIBILITY:
Inclusion Criteria:

* students and teachers in the enrolled schools

Exclusion Criteria:

* students and teachers not enrolled in the schools
* students who did not provide consent or assent to take part in the study

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 9000 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to the PPASF programme's components in the schools | up to 9 months
  Customized fidelity check list based on the 17 program elements.

SECONDARY OUTCOMES:
Number of participants in designated areas of school assessed through a modified version of the SOPLAY protocol | up to 9 months
  A modified version of the "System for Observing Play and Leisure Active In Youth (SOPLAY)" protocol in pre-specified designed areas of the school grounds. The protocol is carried out once a month, carried out by trained students in the school, with assistance of teachers and researchers. Trained students scan the designed area of the school ground from left to right and tally the number of people they encounter that are sedentary, walking or very active. Additional information is collected about the accessibility of the area, the suitability for physical activity, whether there is staff supervision in the area, if the activities are organized physical activity, and if there is any equipment. The count data is marked for each observation period and monitored over time.
Changes in physical activity opportunities through questionnaires | up to 9 months
  Survey items to state the opportunities in school lessons, recess and after-school activities. A check box of sport and physical activities is counted and compared between time points.
Changes in physical activity levels by accelerometer | up to 9 months
  Accelerometers placed on the thigh for a minimum of 4 days (1 weekend day) and at least 10h of wear time per day
Changes in physical activity levels by self-reported physical activity through questionnaires | up to 9 months
  Self-report PA by questionnaire. Two short measures (Prochaska et al, 2001). Both response scales are from 0-7days. Q1 based on the past 7 days. Q2 is based on the average week. Results are averaged and rounded up.
Changes in (accelerometer based) sedentary time during the school day | up to 9 months
  Accelerometers placed on the thigh to measure inclination and algorithm to detect sitting and lying time.
Changes to self-reported academic performance | up to 9 months
  Self-report surveys of perceived academic performance. A four point scale of 'below average' 'average' 'good', 'excellent'.
Changes to self-reported academic performance behaviours | up to 9 months
  Self-report surveys of Harter's self-perception scale for adolescents. Only the Scholastic Competence domain items are used through a structured alternative format. Items grouped into the subscale of Scholastic competence in accordance to the master list of items to produce a summed score.
Changes to school records of Academic behaviours | up to 9 months
  School records of behavours, including absences and behavioural sanctions at the school level, in comparison to previous 5 years records.
Changes in BMI | up to 9 months
  Weight measured in kilograms and height in meters to combine to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Woods, PhD, Principal Investigator — University of Limerick
Locations (1):
- University of Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: January 2020
Access Criteria: By request via the Principal Investigator
URL: https://osf.io/frx6t/

REFERENCES:
- See also: Open Science Framework Link — https://osf.io/frx6t/